CLINICAL TRIAL: NCT03522610
Title: Effectiveness of a Web-enhanced Parenting Program for Military Families
Acronym: ADAPT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1005S82692
Record Dates: First submitted 2018-02-16; First posted 2018-05-11 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Parenting
Keywords: Prevention; Military Families; Parenting

STUDY DESIGN:
Intervention Model Description: This study is a two-group randomized controlled effectiveness trial with baseline and three follow-up assessment points
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ADAPT (Experimental): Parents participate in a 14-week in person group based version of ADAPT with web-enhanced online ADAPT materials.
  Interventions: Behavioral: ADAPT
- Comparison Group (No Intervention): Parents receive services as usual (pamphlets, brochures, etc) on parenting typically found at a VA or Dr.'s office.

INTERVENTIONS:
Behavioral: ADAPT — Two hour, once a week in-person parenting program for 14 weeks plus use web-enhanced supplemental ADAPT materials
  Arms: ADAPT

SUMMARY:
The proposed project will produce and test the first combined group-online prevention program for reintegrating parents - "ADAPT: After Deployment Adaptive Parenting Tools". We will conduct a randomized effectiveness trial of the program, compared with a 'services as usual' (tip sheet) comparison group among 400 military families identified in the RFA as a special population: reintegrating Army National Guard parents.

DETAILED DESCRIPTION:
Combat deployment and related challenges are family stressors, associated with more negative parent-child interactions, ineffective and coercive parenting practices and lower levels of parenting satisfaction. Disrupted parenting practices are well-known predictors of risk for child adjustment difficulties that are precursors to youth substance use, including behavior problems, school failure, deviant peer association, and depression . These child adjustment problems can contribute to continuing parental stress, increasing parental distress, and further disrupting parenting. Despite this, no parenting interventions have been empirically tested for reintegrating military families deployed to OEF/OIF.

PMTO is a well-established empirically supported intervention targeting highly stressed parents that applies Social Interaction Learning theory. Similar to family stress and stress amplification models, SIL posits that parenting mediates the effects of family stressors on child adjustment. That is, deployment and related stressors would be expected to impair social interactional patterns, leading to increases in coercion, decrements in positive parenting, and increased risk for child maladjustment. PMTO interventions have demonstrated efficacy and effectiveness, showing benefits for children including reductions in behavior problems that are precursors to substance use, actual substance use, and internalizing problems, as well as increases in social competence and school adjustment. Moreover, recent findings indicate that strengthening parenting practices contributes to improved outcomes for parents themselves. While PMTO interventions have been implemented in multiple diverse contexts, no study to date has adapted and examined PMTO among military populations. Data from studies of the current wars demonstrate a strong need for accessible prevention interventions that reduce parent stress, enhance parenting, and promote family resilience.

Specific aims of this study are as follows:

1. Examine the usability and feasibility of an adapted PMTO prevention program: After Deployment: Adaptive Parenting Tools/ADAPT

   1. Conduct in-house testing and external usability evaluation of ADAPT online enhancement
   2. Evaluate feasibility of ADAPT group component
2. Assess effectiveness of and satisfaction with ADAPT (group and web enhancement) program compared with a services-as-usual comparison group, among 400 reintegrating MN Army National Guard (MN ARNG) families with 6-12 year old children.

   1. Assess effectiveness of ADAPT in (i) reducing coercion, and improving positive parenting practices, (ii) reducing child risk for substance use and related behavior problems, and (iii) improving parental adjustment, in the face of deployment and reintegration stressors.
   2. Assess the capacity of ADAPT to yield higher parent satisfaction ratings than the services as-usual (tip sheet) comparison condition.
3. Within the ADAPT intervention group, detail and describe responsiveness to intervention.

   1. Report dosage for group (face-to-face) and web components of ADAPT
   2. Examine dosage as a potential moderator of intervention outcome
   3. Examine fidelity of the implementation as a potential moderator of intervention outcome

ELIGIBILITY:
Inclusion Criteria:

1. one parent has returned from deployment to OIF or OEF,
2. at least one child in grades preK-6 in their custody and living with parent(s) in the home, and
3. high speed internet access at home (a recent MN study indicates that 97% deployed families have internet, with 70% using internet daily; Sayer et al., 2009). We will include both single-and two-parent families, as well as families where care is shared between non-partnered adults (e.g. grandparent and mother), and will control for relationship status in analyses. Participants must live within an hour's travel time of the Twin Cities Metro area, St Cloud, Mankato, Duluth, agree to randomization, and indicate willingness to interact with study materials and complete assessment batteries.

Exclusion Criteria:

1. active psychosis,
2. an open child protection case for abuse or neglect in the family,
3. a serious child mental health diagnosis,
4. families who participated in the pilot ADAPT intervention (usability or feasibility) study described in Aim 1. MN NG data indicate that fewer than 10% families would be excluded based on a-c, above (personal correspondence, Polusny).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2010-07-15 (Actual); Primary Completion 2015-07-15 (Actual); Study Completion 2016-07-15 (Actual)

PRIMARY OUTCOMES:
Assess effectiveness of the After Deployment: Adaptive Parenting Tools/ADAPT program | Change from Baseline, at 6 months , at 12 months , at 24 months
  Compare child adjustment with parental adjustment

SECONDARY OUTCOMES:
Examine dosage and participation in ADAPT. | Change from Baseline, at 6 months, at 12 months, at 24 months
  Report dosage for group (face-to-face) vs web components of ADAPT

CONTACTS AND LOCATIONS:
Overall Officials: Abigail Gewirtz, PhD, Principal Investigator — University of Minnesota

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gewirtz AH, DeGarmo DS, Lee S. What works better? 1-year outcomes of an effectiveness trial comparing online, telehealth, and group-based formats of a military parenting program. J Consult Clin Psychol. 2024 May;92(5):310-319. doi: 10.1037/ccp0000882. Epub 2024 Mar 28. PMID 38546621
- [Derived] DeGarmo DS, Gewirtz AH, Li L, Tavalire HF, Cicchetti D. The ADAPT Parenting Intervention Benefits Combat Exposed Fathers Genetically Susceptible to Problem Drinking. Prev Sci. 2023 Jan;24(1):150-160. doi: 10.1007/s11121-022-01424-x. Epub 2022 Sep 3. PMID 36057024
- See also: Current ADAPT studies and history of research — http://adapt.umn.edu